CLINICAL TRIAL: NCT02397343
Title: The Effect of Hyperbaric Oxygen Therapy on Inflammatory Parameters Induced by a Heat Injury Model
Acronym: HBO-SHA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ole Hyldegaard, Consultant, Ass.prof, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HBO-SHA
Record Dates: First submitted 2015-01-22; First posted 2015-03-24 (Estimated); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Secondary Hyperalgesia; Inflammation
Keywords: Reduction of secondary hyperalgesia and/-or local inflammation
MeSH Terms: conditions — Hyperalgesia; Inflammation | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Session 1 (Other): HBO given the first day of study period and sensory test battery performed. 4 weeks later no intervention is given but the sensory test battery performed.
  Interventions: Drug: Hyperbaric oxygen
- Session 2 (Other): No intervention first day of study period and sensory test battery performed. 4 weeks later HBO intervention is given and the sensory test battery performed.
  Interventions: Drug: Hyperbaric oxygen

INTERVENTIONS:
Drug: Hyperbaric oxygen

SUMMARY:
Hyperbaric oxygen may reduce neurophatic pain and promote wound healing. Established anti inflammatory effects of HBO may contribute to this effect. In a previous publication the investigators studied the effects of HBO on secondary hyperalgesia using a well established heat injury model. In a new - blinded study design, the investigators wish to investigate and- or confirm previous results, i.e. that HBO therapy reduce secondary hyperalgesia and improving therapy of severe pain conditions.

DETAILED DESCRIPTION:
Hyperbaric oxygen (HBO) reduces neuropathic pain, promote healing of hypoxic, chronic wounds and sores caused by radiation therapy. Nitric oxide (NO) is a contributing factor to the prolonged anti-nociceptive effect of HBO treatment. In addition, HBO stimulates the formation of reactive oxygen and nitrogen forms, reduces beta-2 integrin function, and reduces contact of leukocytes to the endothelial surface of the capillaries, improves microcirculation and causes decreased monocyte chemokine synthesis. It is the interaction of these mechanisms involved in HBO's anti-inflammatory effect. How HBO reduces pain and inflammation in humans has not been established. In healthy subjects, investigators have shown that HBO has a reducing effect on the mechanism, which at the level the of spinal cord amplifies the number and and the extension of pain impulses. Subjects who were given HBO therapy initially developed significantly less secondary hyperalgesia than the control group several weeks later by the new heat injury suggesting a protective, preconditioning effect. As in the previous experiment (NCT02025686) preconditioning effects will be assessed by means of measurements of thermal thresholds, pin-prick thresholds, erythema indices and secondary hyperalgesic areas (i.e. area under the curve per minute). Similarly,differences in the sequence of sessions (i.e. first session HBO;second session ambient pressure condition or first session ambient pressure condition;second session HBO) will be analyzed accordingly. In an improved blinded study design investigators will now investigate the effect of HBO treatment using the same cutaneous heat injury model, as in the first study. Investigators expect to finally be able to confirm previous results thereby improving treatment of severe pain conditions.

ELIGIBILITY:
Inclusion Criteria:

* male
* speaks and understands danish language
* understood and signed informed consent before medical examination

Exclusion Criteria:

* younger than 18 years of age
* hypertension
* not able to perform equalization of ears and sinuses
* persons who present with a medical history of previous pneumothorax and/- or who may be considered of increased risk of pneumothorax
* diabetics, epilepsia,asthma
* neurological deficits including cognitive as well as psychomotoric disorders
* claustrophobia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Preconditioning | 4 weeks
  Erythema and edema: DermoLab Combo, Cortex Technology, Hadsund. Pain: Is measured at specific times while the heat injury is being made using a VAS scale from 0-10.
  Hyperalgesia: Weighted pins (PinPrick 8, 16, 32, 64, 128, 256, 512 mN) using Dixon's "up-and-down" method.
  Secondary hyperalgesia: PinPrick, 8 symmetrical lines converging towards the center of the heat injury with 45 degrees difference.
  All parameters are compared within the two sessions to assess preconditioning.
Reduction in secondary hyperalgesia | 4 weeks
  Secondary hyperalgesia: PinPrick, 8 symmetrical lines converging towards the center of the heat injury with 45 degrees difference.

SECONDARY OUTCOMES:
Pain reduction | 4 weeks
  Pain: Is measured at specific times while the heat injury is being made using a VAS scale from 0-10.
  Hyperalgesia: Weighted pins (PinPrick 8, 16, 32, 64, 128, 256, 512 mN) using Dixon's "up-and-down" method.
  Secondary hyperalgesia: PinPrick, 8 symmetrical lines converging towards the center of the heat injury with 45 degrees difference.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Hyldegaard, MD, Ph.D, DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen Ø, Denmark